CLINICAL TRIAL: NCT00117065
Title: Study of Transplant Related Anemia Treated With Aranesp® (STRATA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030139
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Anemia
Keywords: Kidney transplant, Renal transplant; Aranesp®, Darbepoetin alfa; Amgen, Q2W dosing, Q4W dosing
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Aranesp®

SUMMARY:
The purpose of this study was to evaluate Aranesp® administered subcutaneously (SC) to maintain hemoglobin (Hb) levels in renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria: - Subjects who are greater than 6 months post-renal transplant (living or cadaveric) - Using adequate contraceptive precaution, if of childbearing potential - Available for follow-up assessments and dosing visits - Hb concentration less than 11.0 g/dL within 3 months of screening and a hemoglobin concentration less than 11.0 during the screening period Exclusion Criteria: - Expected to initiate dialysis or transplantation or be scheduled for a kidney transplant within 6 months of study start, or have less than 1 year life expectancy - Systemic hematologic disease, myeloma, hemolytic anemia, or malignancy (excluding basal cell carcinoma) - Active systemic or chronic infection - Uncontrolled hypertension defined as diastolic blood pressure greater than 110 mm Hg on 2 separate occasions during the 2 weeks prior to screening - Known hypersensitivity to Aranesp® or any of the product's excipients - Disorders that compromise the ability of the subject to give written informed consent and/or to comply with study procedures - Use of any erythropoietic protein or androgen therapy within the 12 weeks prior to screening - Females who are pregnant or breast-feeding - Currently enrolled in or received treatment in an investigational drug/device trial within the past 30 days - Have previously been enrolled in this study - Recent history (within 12 weeks prior to screening) of severe cardiovascular events, grand mal seizure, dialysis or major surgery - Have received a red blood cell transfusion(s) within 8 weeks prior to screening, or currently have active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Hemoglobin values

SECONDARY OUTCOMES:
SF-36 summary and individual domain scores at week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Bloom RD, Bolin P, Gandra SR, Scarlata D, Petersen J. Impact on health-related quality of life in kidney transplant recipients with late posttransplant anemia administered darbepoetin alfa: results from the STRATA study. Transplant Proc. 2011 Jun;43(5):1593-600. doi: 10.1016/j.transproceed.2011.02.009. PMID 21693239
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_200301391.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/